CLINICAL TRIAL: NCT02353507
Title: A Multi-Center, Randomized, Comparison Study of a Chitosan (Opticell Ag+) Silver Dressing and a Sodium Carboxymethylcellulose (Aquacel® Ag+) Silver Dressing on Burn Wounds in Pediatrics and Adults Subjects
Brief Title: Comparison of Chitosan and Carboxymethylcellulose Silver Dressings on Burn Wounds in Pediatric and Adult Subjects
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R14-054
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2015-02

CONDITIONS: Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opticell Ag+ (Active Comparator): Absorbent, antibacterial, barrier dressing
  Interventions: Device: Opticell Ag+
- Aquacel Ag+ (Active Comparator): Absorbent, antibacterial, barrier dressing
  Interventions: Device: Aquacel Ag+

INTERVENTIONS:
Device: Opticell Ag+
  Arms: Opticell Ag+
Device: Aquacel Ag+
  Arms: Aquacel Ag+

SUMMARY:
The purpose of this prospective, randomized, comparative multi-center study is to compare the effective management of two silver-based dressings in managing exudative wounds in first and second degree burns.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient status at the site
* Written consent obtained from the subject
* Burn injury must have been incurred within 36 hours prior to enrollment.
* Burn injury must be of superficial partial thickness, mid-dermal partial thickness, or a combination of the two depths
* Burn injury must exceed 3% total body surface area.

Exclusion Criteria:

* Subject is pregnant.
* Bone fractures.
* Inhalation-related trauma.
* Sensitive and/or allergic to materials containing silver.
* Burn injury exceeds 40% total body surface area.
* Burn injury diagnosis indicates deep partial or full thickness wounds.
* Burn a result of electrical/chemical injury or frostbite.
* An active agent, such as a topical antimicrobial or an enzymatic debriding agent was previously used to treat the burn injury in question.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Wound Infection Rates | Up to 21 days of use
Days required for wound healing | Up to 21 days of use

SECONDARY OUTCOMES:
Pain Levels during Dressing Removal | Up to 21 days
  Categorical scale of pain reported by Subject